CLINICAL TRIAL: NCT00917722
Title: Deep Brain Stimulation of the STN and Cognitive Control: A Pilot Study
Brief Title: Deep Brain Stimulation of the Subthalamic Nucleus (STN) and Cognitive Control
Acronym: COVOLT
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 04-0045
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; STN DBS; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, the investigators will follow patients who have had stimulators implanted, at their usual clinic follow-up appointments 3, 6, 9 and 12 months after surgery. It is typical at these appointments for patients to be off medication and for the stimulators to be turned off to observe disease progress and test stimulator effectiveness. Also as part of standard clinical practice, stimulator settings are adjusted for optimal benefit to motor symptoms. Only patients who already have implants will be invited to participate in this study, and no changes to stimulator settings are made for the purposes of this study. Stimulator settings are changed based on clinical evaluation of motor symptoms, and this study has no bearing on how stimulators will be set nor how often they will be set.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for "definite" Parkinson's Disease (PD)
* STN stimulators on both sides (right and left)
* Surgery done at Washington University within 2 years

Exclusion Criteria:

* Significant visual deficits (e.g. double vision, untreated eyelid apraxia, blepharospasm) Must be able to see screen
* Secondary Parkinsonism (drug-induced or other known etiologies)
* Brain injury or defect: history of serious head injury, stroke, encephalitis, defect found on brain imaging
* Early severe dementia (within first year of onset) or on cholinesterase inhibitors
* Pre-surgical Mini Mental Status exam score < 24
* Significant current psychiatric diagnoses (such as depression or psychosis) or on neuroleptics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Only patients who already have implants will be invited to participate in this study, and no changes to stimulator settings are made for the purposes of this study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara G Hershey, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This was a small pilot study and consent was not obtained to share data.